CLINICAL TRIAL: NCT02995876
Title: The Clinical Performance of Inlay Zirconia Bridges Using Three Different Designs
Brief Title: The Clinical Performance of Inlay Zirconia Bridges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UDDS-FixPro-02-2016
Record Dates: First submitted 2016-12-14; First posted 2016-12-19 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Dental Crowns

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Zirconia and E-max Press (No Intervention): The first design is going to be fabricated with CAD/CAM Zirconia and the occlusal surface from E-max Press.
- Zirconia and E-max Press and Glaze (Experimental): The second design is going to be fabricated with CAD/CAM Zirconia and the occlusal surface from E-max Press and the internal surface coated with a glaze layer to improve adhesion.
  Interventions: Procedure: Glaze layer
- Zirconia and E-max Press twice (Experimental): The third design is going to be fabricated with CAD/CAM Zirconia and the occlusal surface from E-max Press and the internal surface coated with an E-max Press layer to improve adhesion.
  Interventions: Procedure: E-max Press layer

INTERVENTIONS:
Procedure: Glaze layer — A coating of a glaze layer will be used at the inner surface of the bridge to improve adhesion
  Arms: Zirconia and E-max Press and Glaze
Procedure: E-max Press layer — A coating of E-max Press layer will be used at the inner surface of the bridge to improve adhesion
  Arms: Zirconia and E-max Press twice

SUMMARY:
When missing tooth structure or teeth are replaced, minimal biologic risk should be involved to re-establish function and esthetics. The increased use of the adhesive technique and preservation of dental tissues have greatly impacted conservative tooth preparation design. The development use of zirconia technology and all-ceramic systems has opened the potential for fabrication inlays zirconia bridges with durability and good aesthetics.

The purpose of this study is to clinically evaluate the placement of inlay bridge made of a Y-TZP framework veneered with a pressed ceramic and bonded with a completely adhesive approach in the replacement of a single missing tooth.

DETAILED DESCRIPTION:
This study evaluates the use of inlay bridge made of Zirconia and all ceramic systems with three designs in the replacement process of one single tooth (i.e. a missing premolar or molar.) The first design is going to be fabricated with CAD/CAM Zirconia and the occlusal surface from e-max press.

The second design is going to be fabricated with CAD/CAM Zirconia and the occlusal surface from e-max press and the internal surface coated with glaze layer to improve the adhesion.

The third design is going to be fabricated with CAD/CAM Zirconia and the occlusal surface from e-max press and the internal surface coated with a layer of e-max ceramic press to improve the adhesion.

ELIGIBILITY:
Inclusion Criteria:

1. Good oral hygiene
2. Low susceptibility to caries
3. Parallel alignment of abutment teeth
4. Immobility of the abutment teeth
5. Minimum height of abutment teeth ≥ 5 mm (connector thickness)
6. Maximum mesio-distal extension of the inter-dental gap of 9 mm (width of premolar) or 12 mm (width of molar)

Exclusion Criteria:

* Severe para-functional habits.
* Short clinical crowns (<5 mm)
* Extensive defects of the clinical crown,
* Loosening of teeth because of factors related to the periodontal tissues.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Change in marginal fit | Immediately within five minutes following cementation (T1), 3 months (T2), 6 months (T3), 12 months (T4) following application
  To examine if there is a gap between inlay margins and tooth cavity margins .It will be measured by a probe.
Change in Material Integrity | Immediately within five minutes following cementation (T1), 3 months (T2), 6 months (T3), 12 months (T4) following application
  To examine macroscopically the presence of cracks or fractures in the veneering ceramic (retainers or pontics) or any fractures at the connectors.
Change in the Retention Status | Immediately within five minutes following cementation (T1), 3 months (T2), 6 months (T3), 12 months (T4) following application
  The resistance of a prosthesis to displacement will be measured.

SECONDARY OUTCOMES:
Change in Marginal Color Matching | Immediately within five minutes following cementation (T1), 3 months (T2), 6 months (T3), 12 months (T4) following application
  Examination will be done macroscopically to detect the presence of any difference in color between the margins of the tooth and inlays

OTHER OUTCOMES:
Change in Sensitivity | Immediately within five minutes following cementation (T1), 3 months (T2), 6 months (T3), 12 months (T4) following application
  The presence of any spontaneous or stimulated pain will be assumed.
Change in Patients' Satisfaction | Immediately within five minutes following cementation (T1), 3 months (T2), 6 months (T3), 12 months (T4) following application
  A questionnaire will be used to detect the level of satisfaction regarding function and shade
Change in Shade | Immediately within five minutes following cementation (T1), 3 months (T2), 6 months (T3), 12 months (T4) following application
  The shade is going to be determined using Vita(R) shade guide.

CONTACTS AND LOCATIONS:
Overall Officials: Mansour Abo Alkasab, DDS MSc, Principal Investigator — PhD student in Fixed Prosthodontics, University of Damascus Dental School, Damascus, Syria; Jihad Abo Nassar, DDS MSc PhD, Study Director — Associate Professor of Fixed Prosthodontics, University of Damascus Dental School, Damascus, Syria
Locations (1):
- Department of Fixed Prosthodontics, University of Damascus Dental School, Damascus, Syria, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coelho PG, Bonfante EA, Silva NR, Rekow ED, Thompson VP. Laboratory simulation of Y-TZP all-ceramic crown clinical failures. J Dent Res. 2009 Apr;88(4):382-6. doi: 10.1177/0022034509333968. PMID 19407162
- [Background] Cura C, Ozcan M, Isik G, Saracoglu A. Comparison of alternative adhesive cementation concepts for zirconia ceramic: glaze layer vs zirconia primer. J Adhes Dent. 2012 Feb;14(1):75-82. doi: 10.3290/j.jad.a21493. PMID 21594233
- [Background] Monaco C, Ferrari M, Caldari M, Baldissara P, Scotti R. Comparison of 2 bonding systems and survival of fiber-reinforced composite inlay fixed partial dentures. Int J Prosthodont. 2006 Nov-Dec;19(6):577-85. PMID 17165297
- [Background] Raigrodski AJ, Chiche GJ, Potiket N, Hochstedler JL, Mohamed SE, Billiot S, Mercante DE. The efficacy of posterior three-unit zirconium-oxide-based ceramic fixed partial dental prostheses: a prospective clinical pilot study. J Prosthet Dent. 2006 Oct;96(4):237-44. doi: 10.1016/j.prosdent.2006.08.010. PMID 17052467
- [Background] Sanli S, Comlekoglu MD, Comlekoglu E, Sonugelen M, Pamir T, Darvell BW. Influence of surface treatment on the resin-bonding of zirconia. Dent Mater. 2015 Jun;31(6):657-68. doi: 10.1016/j.dental.2015.03.004. Epub 2015 Apr 7. PMID 25862408
- [Background] Valentino TA, Borges GA, Borges LH, Platt JA, Correr-Sobrinho L. Influence of glazed zirconia on dual-cure luting agent bond strength. Oper Dent. 2012 Mar-Apr;37(2):181-7. doi: 10.2341/10-220-L. Epub 2011 Dec 14. PMID 22166107
- [Background] Chaar MS, Kern M. Five-year clinical outcome of posterior zirconia ceramic inlay-retained FDPs with a modified design. J Dent. 2015 Dec;43(12):1411-5. doi: 10.1016/j.jdent.2015.11.001. Epub 2015 Nov 10. PMID 26561926
- [Result] Monaco C, Cardelli P, Ozcan M. Inlay-retained zirconia fixed dental prostheses: modified designs for a completely adhesive approach. J Can Dent Assoc. 2011;77:b86. PMID 21736862